CLINICAL TRIAL: NCT00656357
Title: A Human Laboratory Assessment of the Safety and Potential Efficacy of SYN117 (Nepicastat) in Cocaine-dependent Volunteers Receiving Cocaine
Brief Title: Study of Safety and Potential Efficacy of SYN117 in Cocaine Dependent Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN117-CL01
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-08

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): SYN117 placebo and Ascending doses of cocaine (10, 20, 40 mg) and placebo
  Interventions: Drug: SYN117 Placebo; Drug: Cocaine 10mg; Drug: Cocaine 20mg; Drug: Cocaine 40mg; Drug: Saline
- B (Experimental): Ascending doses of SYN117 (placebo, 80 mg, 160 mg) and ascending doses of cocaine (10 mg, 20 mg, 40 mg) and placebo
  Interventions: Drug: SYN117 80 mg; Drug: SYN117 160 mg; Drug: Cocaine 10mg; Drug: Cocaine 20mg; Drug: Cocaine 40mg; Drug: Saline

INTERVENTIONS:
Drug: SYN117 Placebo — Placebo
  Arms: A
Drug: SYN117 80 mg — SYN117 80 mg
  Arms: B
Drug: SYN117 160 mg — SYN117 160 mg
  Arms: B
Drug: Cocaine 10mg — IV Cocaine 10mg
Drug: Cocaine 20mg — IV Cocaine 20mg
Drug: Cocaine 40mg — IV Cocaine 40mg
Drug: Saline — IV Cocaine Placebo

SUMMARY:
This study will assess the potential interaction and subjective effects between intravenous cocaine and SYN117 in non-treatment seeking cocaine dependant subjects

ELIGIBILITY:
Inclusion Criteria:

* non treatment seeking cocaine dependent
* English speaking
* meet DSM IV TR criteria for cocaine dependence
* pulse 50-90bpm
* systolic BP 85-140 mmHg
* diastolic BP 45-90 mmHg
* essentially normal liver and kidney function blood tests
* ECG normal
* sign informed consent
* negative urine pregnancy test at screening and admission

Exclusion Criteria:

* history or evidence of seizure disorder or brain injury
* previous medically adverse reaction to cocaine, including loss of consciousness, chest pain or epileptic seizure
* neurological disorders, organic brain disease, dementia
* psychiatric disorders such as psychosis, schizophrenia, bipolar disorder, major depression
* history of suicide attempts within past 3 months or suicidal ideation/plan
* history of clinically significant heart disease or hypertension
* family history in 1st degree relatives of early cardiovascular morbidity or mortality
* untreated or unstable medical conditions
* positive HIV test
* pregnant or nursing
* have asthma or are currently using alpha, beta agonists or theophylline or other sympathomimetics
* test positive for other drugs of abuse with the exception of cocaine, cocaine metabolites or marijuana
* any other illness, condition or use of psychotropic medications which preclude safe/successful completion of the study
* currently on parole

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Determine the safety of treatment with SYN117 in cocaine-dependent volunteers by measuring hemodynamic and subjective effects of administration of ascending doses of cocaine(10mg, 20mg, 40mg)and placebo during treatment with ascending doses of SYN117. | inpatient 14 days with 2 week outpatient follow-up

SECONDARY OUTCOMES:
Determine tolerability by measuring adverse events | inpatient 14 days, 2 weeks post followup visit
Determine subjective effects produced by self administration of cocaine or placebo | Days 4, 8, 12 and 13
Determine the effect of SYN117 of the pharmacokinetics of IV cocaine | Days 3 and 11
Determine if any baseline measures of impulsivity or drug use severity predict efficacy of SYN117 in reducing subjective effects of cocaine | Days 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bandak, MD, Study Chair — Biotie Therapies Inc.; F. Gerald Moeller, MD, Study Chair — UTSW-Houston; Kathryn Cunningham, PhD, Principal Investigator — UTMB-Galveston
Locations (1):
- University of Texas Medical Branch (UTMB), Galveston, Texas, United States